CLINICAL TRIAL: NCT07053293
Title: Protocol II: SGLT2i, Hepatic Glucose Production, and Sympathetic Nervous System (SNS)
Brief Title: SGLT2i, Hepatic Glucose Production, and SNS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20230457HU - 504075; R01DK024092 (NIH)
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: Endogenous glucose production; Ketogenesis; Gluconeogenesis; Lipolysis; Norepinephrine turnover
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: A clinical trial comprised of 2 studies
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin (Experimental): Empagliflozin 25 mg/day
  Interventions: Drug: Empagliflozin 25 MG

INTERVENTIONS:
Drug: Empagliflozin 25 MG — A medication used in the management and treatment of type 2 diabetes mellitus. It is in the sodium-glucose co-transporter (SGLT-2) class of medications.
  Other Names: Jardiance

SUMMARY:
In this study, PI will test the hypothesis that distinct mechanisms account for the SGLT2i-induced stimulation of ketogenesis and lipolysis versus endogenous (hepatic) glucose production in patients with type 2 diabetes (T2D) that the increases in ketone production and lipolysis can be prevented by concomitant administration of the thiazolidinedione pioglitazone. Principal Investigator (PI) will conduct five distinct experiments to test this hypothesis in patients with T2D.

To examine the role of the SNS on the empagliflozin-induced stimulation of EGP, lipolysis, and ketone production in T2D by comparing the effect of empagliflozin versus empagliflozin plus propranolol.

DETAILED DESCRIPTION:
Protocol: 22 T2D Subjects will be randomized to receive empagliflozin (n=20). Each subject will participate in two studies performed in random order. In Study 1, EGP will be measured with a prime-continuous 6,6, D2-glucose infusion and lipolysis will be measured with prime-continuous infusion of U-2H-glycerol. The rate of ketogenesis will be determined by infusion of 13C palmitate and quantitating the enrichment of 13C in 3-hydroxybutyrate (BHB). Total body NE turnover will be measured with 3H-norepinephrine (3H-NE) infusion before and after empagliflozin administration.

Visit 2 (Study 1): At approximately 6:00PM on the night prior to study subjects will ingest D2O (3 grams/kg ffm) to quantitate gluconeogenesis and de novo lipogenesis. At 6:00AM at Visit 1 prime-continuous infusions of 6,6, D2-glucose and U-2H-glycerol or U-14C-glycerol are started and continued to study end to measure rates of hepatic glucose production (HGP) and lipolysis. At 8:00AM a prime-continuous infusion of 3H-norepinephrine is started and continued to 9:00 AM at which time it will be stopped. Empagliflozin 25mg is administered at this time, 9:00 AM. At 1:00 PM (240 minutes after administration of Empagliflozin) a second prime-continuous 3H-Norepinephrine infusion is started for 60 minutes. Detailed explanation on page 52-53.

Visit 3 (Study 2, Optional): At approximately 6:00PM on the night prior to study subjects will ingest D2O (3 grams/kg ffm) to quantitate gluconeogenesis and de novo lipogenesis. This visit will be identical to Visit 2 for Aim 2 (Sub-study I) with one exception. At 8:30AM, 30 minutes prior to the ingestion of the Empagliflozin 25mg, a prime (200 ug/kg over 20 minutes)-continuous (80 ug/min) infusion of propranolol is started and continued to study end. Principal Investigator (PI) previously have shown that the steady state propranolol concentration achieved by this infusion rate is sufficient to significantly inhibit insulin-mediated glucose disposal.

ELIGIBILITY:
Patients with T2D

Inclusion Criteria:

* Ages 30-75 years
* Body Mass Index (BMI) 21-45 kg/m2
* Hemoglobin A1C (HbA1c) = 7.0-11%
* Estimated glomerular filtration rate (eGFR) > 60 ml/min/1.73m2
* Blood Pressure (BP) < 160/90 mmHg
* Participants must be in general good health based on medical history, physical exam, screening blood chemistries, complete blood chemistry (CBC), thyroid stimulating hormone/thyroxine (TSH/T4), electrocardiogram (EKG), and urinalysis
* Stable body weight (±1.5 kg) over the last 3 months and must not participate in an excessively heavy exercise program
* Patients treated with diet, sulfonylurea (SU), metformin (MET), or SU/MET
* Statin therapy is permissible if the dose has been stable for at least 3 months

Exclusion Criteria:

* Patients treated with Glucagon-like peptide 1 receptor agonists (GLP-1 RA), Dipeptidyl Peptidase IV inhibitors (DPP-4i), Thiazolidinediones (TZD), or insulin are excluded
* Patients taking medications (other than SU/MET) known to affect glucose metabolism are excluded
* Subjects with evidence of proliferative retinopathy or eGFR < 60 are excluded
* Women of childbearing potential are excluded unless they are taking/using appropriate contractive medications/devices

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Endogenous Glucose Production (EGP) | 0 and 300 minutes
  Measurement of Endogenous Glucose Production (EGP) using stable isotope (6,6, D2- glucose infusion).

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Texas Diabetes Institute/UH, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with NIH and as a publication in a peer reviewed journal once data are published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At study end after analysis of data.